CLINICAL TRIAL: NCT04938843
Title: Effect of F. Prausnitzii on Glycemic Control - a Randomized, Double Blind, Placebo-controlled Study
Brief Title: Effect of F. Prausnitzii on Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MetaboGen AB (Industry)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: META003
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Pre Diabetes; Impaired Glucose Tolerance; Non-Alcoholic Fatty Liver Disease
Keywords: Faecalibacterium prausnitzii; Desulfovibrio piger
MeSH Terms: conditions — Glucose Intolerance; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F. prausnitzii and D. piger (Experimental): 1 capsule administered once daily 45 minutes before breakfast for 12 weeks
  Interventions: Dietary Supplement: F. prausnitzii and D. piger
- Placebo (Placebo Comparator): 1 capsule administered once daily 45 minutes before breakfast for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: F. prausnitzii and D. piger — Dietary supplementation with capsules containing F. prausnitzii and D. piger once daily for 12 consecutive weeks
  Arms: F. prausnitzii and D. piger
Dietary Supplement: Placebo — Dietary supplementation with placebo capsules identical to those containing F. prausnitzii and D. piger once daily for 12 consecutive weeks
  Arms: Placebo

SUMMARY:
The microbiota is associated with a wide spectrum of diseases including diabetes and non-alcoholic fatty liver disease. In this study we will investigate if the bacteria F. prausnitzii, which is a part of the human gut microbiota, can improve metabolic parameters in subjects with impaired glucose control.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled study. Subjects with impaired glucose control will after signing the informed consent and fulfilling the study criteria be randomized to study product or placebo. The randomization ratio between the study product (F. prausnitzii 1E8-5x1E8 CFU and D. piger) and placebo is 1:1. In total 176 subjects will be randomized in the study.

The study will start with a Run-in period i.e. all the subjects will be given placebo capsules. The subjects fulfilling the inclusion and exclusion criteria will be randomized at Visit 2 to either study product or placebo in the ration 1:1. The treatment will last for 12 weeks, from Visit 2 to Visit 6. The study is ended with a 2-week period of follow up after the final dose.

Blood samples are taken at Visits 1-4 and Visits 6-7. Feces samples are collected at Visit 2-7. One additional fecal sample will be sent by mail approximately one week after Visit 1. Glucose monitoring (CGM) will be initiated at Visit 1 and Visit 5 and followed for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Man or woman 50-75 years of age
* Impaired glucose tolerance (IGT; capillary b-glucose 8.9-12.1 mmol/L, 120 minutes after OGTT), impaired fasting glucose (IFG; capillary b-glucose 6.1-6.9 mmol/L) or combined glucose intolerance (CGI, i.e. IFG and IGT)
* Weight stable ±5 kg for the last 3 months, BMI >18 kg/m2
* Willingness and possibility to come to the planned study visits, use the Diary and eQuestionnaires as well as follow the study instructions
* Understand Swedish in speech and writing

Exclusion Criteria:

* Other reasons for liver inflammation e.g. hepatitis A, hepatitis B, hepatitis C, HIV-positive, confirmed or suspected cirrhosis, Wilsons disease, autoimmune hepatitis, hemochromatosis, alcohol related fatty liver or pancreatitis, laboratory screen AST/ALT >2 (ULN), Bilirubin >1 (ULN)
* Heart failure NYHA class III, cardiovascular event within 6 months, unstable angina pectoris
* Diabetes mellitus, HbA1c >47 mmol/mol or fp-Glucose >6.9 mmol/L on 2 occasions
* Chronic obstructive pulmonary disease and asthma treated with intermittent steroids to be under control
* Blood pressure >170/105 mmHg
* Blood donation >500 mL blood <3 months before screening
* Anemia, Hb <117 g/L females and Hb <134 g/L males; leukopenia, LPK <3.5x1E9/L, ongoing infection CRP >10 mg/L
* Hyperthyroidism, T4 >22 nmol/L or hypothyroidism, TSH >4,2 mIU/L
* Laboratory result of clinical significance meaning that participation in the study is unsuitable according to Investigator
* Calculated glomerular filtration rate (GFR) <60 mL/min/1.73 m2
* Cancer <5 years since diagnosis, except for basal-cell carcinoma
* Treatment during the last 3 months with oral steroids, biological drugs, immunosuppressive drugs, e.g. cyklosporin, drugs known to cause liver damage or to be liver toxic
* Bariatric surgery
* Antibiotic treatment during the last 3 months or reoccurring antibiotic treatment >3 times a year
* Regular or sporadic use of probiotic product (not food containing probiotics) during the last 3 months
* Confirmed IBD, irritable bowel syndrome (IBS), bile acid malabsorption, gastrointestinal infections during the last 3 months or any experienced problems from the gastrointestinal tract during the last month that the Investigator expect could influence the participation in the study
* Allergy to metronidazol, the adhesive glue for the CGM sensor, milk protein
* Smoking >10 cigarettes/day
* Alcohol consumption, >7 units/week females, >14 units/week males
* Use of narcotics e.g. cannabis, amphetamine (not medical use), hallucinogens, gamma-hydroxybutyric acid
* Pregnancy, breast-feeding or planned pregnancy
* Participation in other studies except IGT2

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | From baseline to week 12
  Change in time (%) glucose concentration range of 3.5-6.0 mmol/L measured with continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Fasting plasma glucose levels | From baseline to week 12
  Change in fp-glucose
Hemoglobin A1c | From baseline to week 12
  Change in b-HbA1c
Homeostatic Model Assessment (HOMA) for Insulin Resistance (IR) | From baseline to week 12
  Change in HOMA-IR
Continuous glucose monitoring (CGM) mean | From baseline to week 12
  Change in CGM mean
CGM SD | From baseline to week 12
  Change in CGM SD
CGM CV | From baseline to week 12
  Change in CGM CV
CGM MAGE | From baseline to week 12
  Change in CGM MAGE
Glucose levels | From baseline to week 12
  Change in CGM time (%) glucose concentration ≥7.0 mmol/L
Liver fat content | From baseline to week 12
  Change in liver fat measured by transient elastography and given as CAP (continous attenuation parameter) in db/m
Liver fat content | From baseline to week 12
  Change in liver fat measured by ultrasound (kPa)
Liver fat function test AST | From baseline to week 12
  Change in AST
Liver fat function test ALT | From baseline to week 12
  Change in ALT
Liver fat function test GGT | From baseline to week 12
  Change in GGT

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, Principal Investigator — Wallenberg Laborotory, University of Gothenburg
Locations (1):
- Wallenberg Laboratory, University of Gothenburg, Gothenburg, Västra Götaland County, Sweden